CLINICAL TRIAL: NCT05061199
Title: The Impact of Intracorporeal Anastomosis on Resection Margin During Laparoscopic Radical Resection of Transverse Colon Cancer: a Retrospective Multi-center Study
Brief Title: Resection Margin of Transverse Colon Cancer With Extracorporeal Versus Intracorporeal Anastomosis
Status: Completed | Type: Observational
Sponsor: Shanghai Minimally Invasive Surgery Center (Other)
Responsible Party: Sponsor
Other Study IDs: MISC-TCC-ECA-ICA
Record Dates: First submitted 2021-09-18; First posted 2021-09-29 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Transverse Colon Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ECA group: TCC with extracorporeal anastomosis (ECA)
  Interventions: Procedure: approach of anastomosis
- ICA group: TCC with intracorporeal anastomosis (ICA).
  Interventions: Procedure: approach of anastomosis

INTERVENTIONS:
Procedure: approach of anastomosis — The approach of anastomosis

SUMMARY:
The approach of anastomosis in laparoscopic resection of transverse colon cancer (TCC) has rarely been discussed. This study aims to compare the resection margin of TCC with extracorporeal anastomosis (ECA) versus intracorporeal anastomosis (ICA).

Patients who underwent laparoscopic resection of TCC from August 2019 to July 2021 in 13 participating centers are included in this study. According to the approach of anastomosis, patients are divided into two groups, ECA group and ICA group respectively. The clinical characteristics, the perioperative outcomes and the pathological results (especially the length of resection margin) are compared between the two groups. The length of two-sided resection margins (long margin, short margin) are measured on formalin-fixed specimens and those with short margin less than 4.0 cm are defined as unqualified specimens.

DETAILED DESCRIPTION:
13 participating centers are as follows: Ruijin Hospital, Shanghai Jiaotong University School of Medicine；Zhejiang University Medical College Affiliated Sir Run Shaw Hospital；Zhongshan Hospital Affiliated to Fudan University；Renji Hospital Affiliated to Medical College of Shanghai Jiaotong University; Jiangsu Provincial People's Hospital; Xiangya Hospital of Central South University; The First Affiliated Hospital of Chongqing Medical University; The first hospital of Jilin University; Beijing Friendship Hospital Affiliated to Capital Medical University; Tangdu Hospital; Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of science and technology; Cancer Hospital of Chinese Academy of Medical Sciences; Henan Provincial People's Hospital

ELIGIBILITY:
Inclusion Criteria:

* 1. pathologically confirmed adenocarcinoma of colon
* 2. The tumor is located in the transverse colon (including hepatic or splenic flexure);
* 3. One of the following procedures was performed: transverse colectomy, right hemicolectomy, enlarged right hemicolectomy, left colectomy, enlarged left colectomy;
* 4. Laparoscopic surgery (laparoscopy-assisted surgery or complete laparoscopic surgery) from August 2019 to July 2021;
* 5. Radical resection (R0) was accomplished;

Exclusion Criteria:

* 1. Simultaneous multiple colorectal cancer;
* 2. history of colorectal surgery (except endoscopic surgery);
* 3. robot-assisted surgery;
* 4. palliative resection (non-R0 resection) or palliative bypass;
* 5. the approach of anastomosis could not be determined from the documents;
* 6. the length of resection margin was not recorded in pathological report;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: transverse colon cancer
Sampling Method: Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
length of the resection margin | one month after surgery
  length of the two -sided resection margins measured on formalin-fixed specimen (CM)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Minimally Invasive Surgery Center, Shanghai, China

REFERENCES:
- [Derived] Zhong H, Cai Z, Lu J, Yang Y, Xu Q, Wang N, He L, Hu X, Fingerhut A, Zheng M, Lu A, Liu Z, Xiao Y, Feng B. Pathological and perioperative outcomes of extracorporeal versus intracorporeal anastomosis in laparoscopic transverse colon cancer resection: retrospective multicentre study. BJS Open. 2023 May 5;7(3):zrad045. doi: 10.1093/bjsopen/zrad045. PMID 37161672